CLINICAL TRIAL: NCT02184676
Title: Early Immunological, Metagenomic, Metabolic and Environmental Factors in the Progression to Type 1 Diabetes: the TRAKR Cohort
Brief Title: T1D Risk Assessment in Kids With Relatives
Acronym: TRAKR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé et de la Recherche Médicale (INSERM) U1016 - Institut Cochin, Immunology of Diabetes Team, Paris, France (Unknown); INSERM U1153, Epidemiology Research Unit on Perinatal Health and Women and Children Health, Port-Royal Hospital, Paris, France (Unknown); Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other); Commissariat A L'energie Atomique (Other Government); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: P130405; ID RCB : 2014-A00453-44
Record Dates: First submitted 2014-07-03; First posted 2014-07-09 (Estimated); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; risk assessment; immunological marker; children; relatives; autoantibodies; lymphocytes; T cells; epitopes; Children born to mother/father with type 1 diabetes and their parents
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Children born to mother/father with type 1 diabetes (Other)
  Interventions: Biological: Analysis of early immune modifications; Other: Collection of clinical and socio-demographic data

INTERVENTIONS:
Biological: Analysis of early immune modifications — * blood and stool sampling in parents during pregnancy (at enrollment, i.e. 7th-8th month of pregnancy)
  * cord blood sampling
  * stool sampling in mothers and newborns at birth (day 7)
  * blood and stool sampling in children at the age of 8, 18, 30 and 42 months
Other: Collection of clinical and socio-demographic data — 1. Questionnaire filled in by clinicians at enrollment and at birth
  2. Self-administered questionnaire filled by parents at enrollment, at birth, and then at month 8, 18, 30 and 42

SUMMARY:
The purpose of this study is to determine whether early immunological markers (activation of autoreactive T lymphocytes) precede and are predictive of the appearance of autoantibodies in children born from type 1 diabetic parents.

DETAILED DESCRIPTION:
The prevalence of type 1 diabetes (T1D) is estimated between 0.2 and 0.4% in France. The incidence in France is more than 10/105 per year, with a steady increase (~4%/year), especially in children. Infants born to parents with T1D have a 15-fold higher risk to develop T1D compared to the general population. The appearance of autoantibodies precedes and is highly predictive of the later occurrence of T1D. The activation of B lymphocytes, which produce autoantibodies, is controlled by T helper lymphocytes. Hence, biomarkers associated with initial T lymphocyte activation are likely to precede the appearance of autoantibodies.

The aim of the TRAKR study is to determine whether the appearance of autoreactive T lymphocytes is predictive of the emergence of autoantibodies.

The secondary objectives are: 1) to evaluate whether metagenomic, metabolic, or environmental factors are associated with the appearance of autoantibodies; 2) to evaluate the incidence and the time of autoantibody appearance in a French population of genetically at-risk children; 3) to compare the incidence of autoantibodies between infants born to T1D fathers and mothers.

ELIGIBILITY:
Inclusion Criteria:

1. Mother and/or father with type 1 diabetes

   * age > 18 years
   * type 1 diabetes : insulin-dependent diabetes positive for autoantibodies against insulin and/or GAD and/or IA-2 and/or ZnT8 at the time of diagnosis
   * planning to give birth or having given birth since less than 8 months
   * agreeing to participate upon written informed consent
   * covered by the French social security system
2. Mother/father without Type 1 diabetes

   * age > 18 years old
   * with a spouse with type 1 diabetes : insulin-dependent diabetes positive for autoantibodies against insulin and/or GAD and/or IA-2 and/or ZnT8 at the time of diagnosis
   * planning to give birth or having given birth since less than 8 months
   * agreeing to participate upon written informed consent
   * covered by the French social security system
3. Children born to mother and/or father with type 1 diabetes

   * age < 8 months
   * with at least one parent with T1D
   * with both parents agreeing to participate
   * both parents covered by the French social security system

Exclusion Criteria:

1) Mother/father

* secondary forms of diabetes
* monogenic forms of diabetes

  1 or 2) For the mother
* malignant neoplastic or psychiatric disease

  3 ) Newborns of mother/father with type 1 diabetes
* Severe foetal disease
* Severe congenital malformation
* Congenital measles

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2015-05-28 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2019-05-17 (Actual)

PRIMARY OUTCOMES:
Autoreactive T lymphocytes | 48 months
  presence, frequency, antigen specificity, phenotype

SECONDARY OUTCOMES:
Metagenomic signatures | 48 months
  presence, frequency, type
Metabolic signatures | 48 months
  presence, frequency, type
Environmental factors | 48 months
  1. Sociodemographic characteristics, e.g. age, gender, occupation, living place, family situation, number of children, education, housing type, animal contact
  2. Family history, e.g. autoimmune diseases
  3. Personal history, e.g. diabetes characteristics, associated co-morbidities, obstetrical history
  4. Clinical data
Incidence of autoantibodies | 48 months
  Presence, titer, specificity

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Mallone, M.D, Ph.D., Principal Investigator — INSERM U1016
Locations (1):
- Cochin Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No